CLINICAL TRIAL: NCT01738269
Title: A Multi-center Reference Value Study of Elecsys HE4 in Chinese Population
Brief Title: Elecsys HE4 Chinese Reference Value Study
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yaping Tian, Director of Biochemistry Department, Chinese PLA General Hospital
Other Study IDs: CIM RD001
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer, HE4, normal range
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Apparently healthy subjects
- Non-malignant conditions subjects
- Malignant conditions subjects

SUMMARY:
Aim of this study is to provide specimens for establishing reference values of HE4 in an apparently healthy Chinese population using the Roche Elecsys HE4 assay tested on variety of Elecsys and cobas brand immunoassay analyzers. This reference range will be compared to population of subjects who have signs and symptoms of various benign and malignant diseases, including ovarian cancer. This reference range will also be compared to the levels of HE4 in individual subjects who have been diagnosed with ovarian cancer and are being followed longitudinally for recurrence or progression of their disease.

ELIGIBILITY:
Inclusion Criteria (all cohorts):

* appropriate clinical data
* normal appearance of sample
* minimum 0.5 ml volume available

Exclusion Criteria (all cohorts):

* < 18 years of age
* insufficient volume
* insufficient clinical information
* > 3 freeze/thaw cycles of samples
* Stored or shipped at > 0°C
* Icteric, lipemic, hemolytic, substantial particulates

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Except for samples from apparently healthy subjects, specimens for the entire clinical section are supposed to be available in banks / archives. Thus, for the most part, no prospective collection of serum should be necessary. Pseudonymized residual samples will be used. All elements of the clinical part require samples from well characterized cohorts are showed below.
  1. Apparently Healthy: 300
  2. Non-malignant Conditions: 650
  3. Malignant Conditions: 800
Sampling Method: Non-Probability Sample
Enrollment: 2351 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Establish reference in Chinese population | October 2012 - March 2013

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - China PLA General Hospital, Beijing
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Sun Yat-Sen University Cancer Center, Guangzhou
  - Shandong University Qilu Hospital, Jinan
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tianjin Cancer Hospital, Tianjin
  - Xinjiang Medical University Cancer Center, Ürümqi
  - Tongji Hospital Tongji Medical Colege of HUST, Wuhan
  - Zhongshan Hospital Xiamen University, Xiamen